CLINICAL TRIAL: NCT05210621
Title: LONG-TERM EFFECTIVENESS AND SAFETY EVALUATION OF OCRELIZUMAB IN FRENCH PATIENTS WITH PROGRESSIVE MS: CONSONANCE EXTENSION STUDY
Brief Title: LONG-TERM EFFECTIVENESS AND SAFETY EVALUATION OF OCRELIZUMAB
Acronym: CONSONANCE EX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-PP-23
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with MS who have completed the CONSONANCE study (Other)
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — ocrelizumab will be administered as single 600-mg infusions in 500 mL 0.9% sodium chloride every 24 weeks (±14 days) up to Week 192 (Year 4) of this study

SUMMARY:
The study duration of 4 years was considered to be sufficient to show a reliable and relevant effect of ocrelizumab on disability progression in the main study (CONSONANCE). However, given the potential long-term use of ocrelizumab in patients with progressive MS, it is critical that additional effectiveness and safety data are accrued in this patient population. In particular, understanding how ocrelizumab can prevent or delay time to major disability milestones such as the need to use an assisting device (Expanded Disability Status Scale [EDSS] 6.0) or a wheelchair (EDSS ≥7.0) is of significant relevance, given that progression to such milestones is associated with a significant reduction in patients' quality of life and an increase in cost of treatment (Kobelt et al. 2017).

In the ORATORIO trial, ocrelizumab reduced the risk of 24-week confirmed EDSS ≥7.0 by 46% (hazard ratio [HR]: 0.54, 95% CI 0.31-0.92; p = 0.022) in patients with primary progressive multiple sclerosis (PPMS). To further characterize the potential long-term impact of ocrelizumab treatment on time to 24-week confirmed EDSS ≥7.0, an analysis was used to extrapolate the observed data into the future, estimating the time at which 50% of patients were expected to have reached EDSS ≥7.0. Extrapolated median time to confirmed EDSS ≥7.0 was 12.1 years for placebo, which was similar to the actual median time observed in MSBase (12.4 years), and 19.2 years for ocrelizumab, representing a 7.1-year delay (95% CI: -4.3 to 18.4) [Butzkueven et al 2021]. A recent MSBase analysis also showed that in a cohort of patients with secondary progressive MS (SPMS), 17.9% reached a confirmed EDSS score of 7.0 from the diagnosis of SPMS, over a period of approximately 12 years (Lizak et al. 2020). Therefore, following patients who complete CONSONANCE beyond the 4-year study period is justified, to better assess the impact of ocrelizumab on these long-term disability milestones.

Another important therapeutic clinical goal in patients with progressive MS is preserving upper limb function. Patients with progressive MS with high EDSS scores, including those who are wheelchair-restricted, experience a devastating reduction in quality of life if they lose any residual function in their arms and/or hands, as this affects the level of independence and significantly limits the ability to perform activities of daily living (Kraft et al. 2014). The Nine-Hole Peg Test (9-HPT) has become one of the most frequently used measures of upper extremity function in MS (Earhart et al. 2011). A 20% worsening in test time is commonly used to define clinically meaningful worsening, as it corresponds to predefined clinically significant changes of established clinician- and patient-reported measures (Feys et al. 2017). Progression rates are lower for 9-HPT compared to EDSS or the Timed 25-Foot Walk Test (25FWT; Goldman et al. 2019). Therefore, following patients who complete CONSONANCE beyond the 4 year study period is justified, to better assess the long-term impact of ocrelizumab on preserving upper limb function.

Patients with MS who have completed the CONSONANCE study, and have a favorable benefit risk ratio, as determined by the treating neurologist, can be included in this study if they meet the inclusion and exclusion criteria.

1.1. Study design

This is a 4-year, single-arm, open-label, multicenter study for patients who have completed 192 weeks of treatment with ocrelizumab in the CONSONANCE study (NCT03523858), and enrolled under the protocol version 1 of CONSONANCE. It is estimated that the study will enroll approximately 90 patients with progressive MS. The study will consist of the following periods:

1. Screening period: The screening visit should be scheduled up to two weeks before the first infusion of ocrelizumab, and always after the last visit of CONSONANCE at Week 192. This period should not be exceeded.
2. Treatment period: The first visit of the treatment period (first infusion of ocrelizumab) will occur at the baseline visit, which should be 24 weeks (+14 days) after the last infusion of ocrelizumab in CONSONANCE. Ocrelizumab will be administered every 24 weeks up to Week 168 of this study. The last visit in the treatment period will be conducted 24 weeks after the last dose of ocrelizumab (i.e., at Week 192).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Able to comply with the study protocol, in the investigator's judgment
* Affiliation to the social security system
* Completed the treatment period of Roche-sponsored ocrelizumab trial (CONSONANCE) and who in the opinion of the investigator may benefit from treatment with ocrelizumab. Only patients enrolled under Protocol version 1 (approval date: 18 February 2018) will be eligible.
* Meet re-treatment criteria with ocrelizumab (please see section 6.11)
* Patients who became pregnant by chance between the last visit of the CONSONANCE study and screening of this study, as confirmed by pregnancy tests at screening, will enter the study but will only re-start treatment with ocrelizumab after birth or after breastfeeding is stopped, as per re-treatment criteria in section 6.11
* Women of childbearing potential* (WOCBP):

  * Must have a negative urine pregnancy test at Visit 1 (Screening) and Visit 2 (Baseline)
  * Must agree to remain abstinent or use an acceptable birth control method during the treatment period and for at least 6 months or longer after the final dose of ocrelizumab, as applicable in the ocrelizumab package leaflet. The following contraceptive methods are considered acceptable (failure rate >1% [Clinical Trial Facilitation Group (CTFG)]): (1) progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action; (2) male or female condom with or without spermicide; (3) cap, diaphragm, or sponge with spermicide; (4) combination of male condom with cap, diaphragm, or sponge with spermicide (double-barrier method). Birth control methods that are highly effective (i.e. failure rate <1% [CTFG]) may also be used but are not required, and include: (1) oral, intravaginal or transdermal combined hormonal contraception associated with inhibition of ovulation; (2) oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; (3) intrauterine device; (4) intrauterine hormone-releasing system; (5) bilateral tubal occlusion; (6) vasectomized partner; (7) sexual abstinence.

Exclusion Criteria:

* Hypersensitivity to ocrelizumab or any of its excipients
* Patients in a severely immunocompromised state, until the condition resolves
* Evidence of any adverse event (AE) potentially attributable to ocrelizumab, for which the local label recommends permanent discontinuation
* Existence of a contra-indication as per the Summary of Product Characteristics (SmPC)
* Prohibited concomitant medication as specified in section 6.7
* Patients intending to become pregnant during the study or within 6 months after the last dose of the study drug in CONSONANCE
* Patients who had early ocrelizumab discontinuation in CONSONANCE (exemption made for treatment discontinuation due to unplanned pregnancy and breastfeeding for patients who continued clinical study assessments in CONSONANCE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2029-02-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with upper limb disability progression | baseline
  Proportion of patients with upper limb disability progression, defined as the proportion of patients with ≥20% worsening in 9 HPT score confirmed for at least 24 weeks,
Proportion of patients with upper limb disability progression | week 192.
  Proportion of patients with upper limb disability progression, defined as the proportion of patients with ≥20% worsening in 9 HPT score confirmed for at least 24 weeks,

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Amiens University Hospital, Amiens
  - Bayonne Hospital, Bayonne
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - Clermont ferrand University Hospital, Clermont-Ferrand
  - Lille University Hospital, Lille
  - Lyon University Hospital, Lyon
  - Marseille Univesity Hospital, Marseille
  - Montpellier University Hospital, Montpellier
  - Nancy University Hospital, Nancy
  - Nantes University hospital, Nantes
  - Nice University Hospital, Nice
  - Nimes University Hospital, Nîmes
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg